CLINICAL TRIAL: NCT02074150
Title: ASIS for Botox in Upper Limb Spasticity
Acronym: ASISinULS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: li nguyen (Industry)
Responsible Party: Sponsor-Investigator, li nguyen, MD/CEO/PI, ASIS Corporation
Organization: ASIS Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCTHD081800; R44HD081800 (Other Grant/Funding Number: EUNICE KENNEDY SHRIVER NATIONAL INSTITUTE OF CHILD HEALTH)
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Upper Limb Spasticity Unilaterally in Adults With History of Stroke; Increased Muscle Tone in Elbow, Wrist, Finger, and Thumb Flexors.
Keywords: Subdermal bloodless space; Subdermal injection; injectable EMG needle; electrical stimulation; MRI with Gadolinium; Upper Limb Spasticity; intramuscular injection
MeSH Terms: interventions — Gadolinium; Gadolinium DTPA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (23):
- Biceps Brachii (Experimental): Biceps Brachii (elbow flexors)
  Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9ccNS intramuscularly for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium
- Flexor Carpi Radialis (Experimental): Flexor Carpi Radialis (wrist flexors)
  Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9ccNS intramuscularly for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium
- Flexor carpi ulnaris (Experimental): Flexor carpi ulnaris (wrist flexors)
  Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9ccNS intramuscularly for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium
- Flexor digitorum profundus (Experimental): Flexor digitorum profundus (finger flexors)
  Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9ccNS intramuscularly for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium
- Flexor digitorum sublimis (Experimental): Flexor digitorum sublimis (finger flexors)
  Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9ccNS intramuscularly for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium
- Adductor pollicis (Experimental): Adductor pollicis (thumb flexors)
  Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9ccNS intramuscularly for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium
- Flexor pollicis longus (Experimental): Flexor pollicis longus (thumb flexors)
  Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9ccNS intramuscularly for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium
- Change from Baseline in Elbow Ashworth (Experimental): Change from Baseline in Elbow Ashworth Scale as Efficacy of Botox intramuscularly at Week 6, Efficacy of Botox intramuscularly at Week 12, Efficacy of Botox intramuscularly at Week 18, Efficacy of Botox intramuscularly at Week 24, and Efficacy of Botox intramuscularly at Week 30 vs.Efficacy of Botox subdermally at Week 6, Efficacy of Botox subdermally at Week 12, Efficacy of Botox subdermally at Week 18, Efficacy of Botox subdermally at Week 24, and Efficacy of Botox subdermally at Week 30. Ashworth score (the force required to move an extremity around a joint):
  0 = No increase in muscle tone (none)
  1. = Slight increase
  2. = Moderate increase
  3. = Considerable increase
  4. = Limb rigid (very severe).
  Interventions: Drug: Efficacy of Botox intramuscularly at Week 6; Drug: Efficacy of Botox intramuscularly at Week 12,; Drug: Efficacy of Botox intramuscularly at Week 18; Drug: Efficacy of Botox intramuscularly at Week 24; Drug: Efficacy of Botox intramuscularly at Week 30; Drug: Efficacy of Botox subdermally at Week 6; Drug: Efficacy of Botox subdermally at Week 12; Drug: Efficacy of Botox subdermally at Week 18; Drug: Efficacy of Botox subdermally at Week 24; Drug: Efficacy of Botox subdermally at Week 30
- Change from Baseline in Wrist Ashworth (Experimental): Change from Baseline in Wrist Ashworth Scale as Efficacy of Botox intramuscularly at Week 6, Efficacy of Botox intramuscularly at Week 12, Efficacy of Botox intramuscularly at Week 18, Efficacy of Botox intramuscularly at Week 24, and Efficacy of Botox intramuscularly at Week 30 vs.Efficacy of Botox subdermally at Week 6, Efficacy of Botox subdermally at Week 12, Efficacy of Botox subdermally at Week 18, Efficacy of Botox subdermally at Week 24, and Efficacy of Botox subdermally at Week 30.Ashworth score (the force required to move an extremity around a joint):
  0 = No increase in muscle tone (none)
  1. = Slight increase
  2. = Moderate increase
  3. = Considerable increase
  4. = Limb rigid (very severe).
  Interventions: Drug: Efficacy of Botox intramuscularly at Week 6; Drug: Efficacy of Botox intramuscularly at Week 12,; Drug: Efficacy of Botox intramuscularly at Week 18; Drug: Efficacy of Botox intramuscularly at Week 24; Drug: Efficacy of Botox intramuscularly at Week 30; Drug: Efficacy of Botox subdermally at Week 6; Drug: Efficacy of Botox subdermally at Week 12; Drug: Efficacy of Botox subdermally at Week 18; Drug: Efficacy of Botox subdermally at Week 24; Drug: Efficacy of Botox subdermally at Week 30
- Change from Baseline in Finger Ashworth (Experimental): Change from Baseline in Finger Ashworth Scale as Efficacy of Botox intramuscularly at Week 6, Efficacy of Botox intramuscularly at Week 12, Efficacy of Botox intramuscularly at Week 18, Efficacy of Botox intramuscularly at Week 24, and Efficacy of Botox intramuscularly at Week 30 vs.Efficacy of Botox subdermally at Week 6, Efficacy of Botox subdermally at Week 12, Efficacy of Botox subdermally at Week 18, Efficacy of Botox subdermally at Week 24, and Efficacy of Botox subdermally at Week 30. Ashworth score (the force required to move an extremity around a joint):
  0 = No increase in muscle tone (none)
  1. = Slight increase
  2. = Moderate increase
  3. = Considerable increase
  4. = Limb rigid (very severe).
  Interventions: Drug: Efficacy of Botox intramuscularly at Week 6; Drug: Efficacy of Botox intramuscularly at Week 12,; Drug: Efficacy of Botox intramuscularly at Week 18; Drug: Efficacy of Botox intramuscularly at Week 24; Drug: Efficacy of Botox intramuscularly at Week 30; Drug: Efficacy of Botox subdermally at Week 6; Drug: Efficacy of Botox subdermally at Week 12; Drug: Efficacy of Botox subdermally at Week 18; Drug: Efficacy of Botox subdermally at Week 24; Drug: Efficacy of Botox subdermally at Week 30
- Change from Baseline in Thumb Ashworth (Experimental): Change from Baseline in Thumb Ashworth Scale as Efficacy of Botox intramuscularly at Week 6, Efficacy of Botox intramuscularly at Week 12, Efficacy of Botox intramuscularly at Week 18, Efficacy of Botox intramuscularly at Week 24, and Efficacy of Botox intramuscularly at Week 30 vs.Efficacy of Botox subdermally at Week 6, Efficacy of Botox subdermally at Week 12, Efficacy of Botox subdermally at Week 18, Efficacy of Botox subdermally at Week 24, and Efficacy of Botox subdermally at Week 30. Ashworth score (the force required to move an extremity around a joint):
  0 = No increase in muscle tone (none)
  1. = Slight increase
  2. = Moderate increase
  3. = Considerable increase
  4. = Limb rigid (very severe).
  Interventions: Drug: Efficacy of Botox intramuscularly at Week 6; Drug: Efficacy of Botox intramuscularly at Week 12,; Drug: Efficacy of Botox intramuscularly at Week 18; Drug: Efficacy of Botox intramuscularly at Week 24; Drug: Efficacy of Botox intramuscularly at Week 30; Drug: Efficacy of Botox subdermally at Week 6; Drug: Efficacy of Botox subdermally at Week 12; Drug: Efficacy of Botox subdermally at Week 18; Drug: Efficacy of Botox subdermally at Week 24; Drug: Efficacy of Botox subdermally at Week 30
- Change from Baseline in PGAS (Experimental): Change from Baseline in PGAS as Efficacy of Botox intramuscularly at Week 6, Efficacy of Botox intramuscularly at Week 12, Efficacy of Botox intramuscularly at Week 18, Efficacy of Botox intramuscularly at Week 24, and Efficacy of Botox intramuscularly at Week 30 vs.Efficacy of Botox subdermally at Week 6, Efficacy of Botox subdermally at Week 12, Efficacy of Botox subdermally at Week 18, Efficacy of Botox subdermally at Week 24, and Efficacy of Botox subdermally at Week 30. The Physician Global Assessment Scale or PGAS is a 9 category scale scoring the physician's evaluation of the patients' status compared to baseline, ranging from -4 to +4 (very marked worsening to complete improvement), with 0 indicating no change from baseline and +1 slight improvement.
  Interventions: Drug: Efficacy of Botox intramuscularly at Week 6; Drug: Efficacy of Botox intramuscularly at Week 12,; Drug: Efficacy of Botox intramuscularly at Week 18; Drug: Efficacy of Botox intramuscularly at Week 24; Drug: Efficacy of Botox intramuscularly at Week 30; Drug: Efficacy of Botox subdermally at Week 6; Drug: Efficacy of Botox subdermally at Week 12; Drug: Efficacy of Botox subdermally at Week 18; Drug: Efficacy of Botox subdermally at Week 24; Drug: Efficacy of Botox subdermally at Week 30
- Adverse Reactions with Facial paresis (Experimental): Facial paresis as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Eyelid ptosis (Experimental): Eyelid ptosis as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Bronchitis (Experimental): Bronchitis as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Neck pain (Experimental): Neck pain as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Muscle stiffness (Experimental): Musculoskeletal stiffness as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Muscular weakness (Experimental): Muscular weakness as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Myalgia (Experimental): Myalgia as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Muscle pain (Experimental): Musculoskeletal pain as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Muscle spasms (Experimental): Muscle spasms as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions Injection site pain (Experimental): Injection site pain as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Hypertension (Experimental): Hypertension as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally

INTERVENTIONS:
Drug: Gadolinium — Gadolinium .1cc/ diluted with .9ccNS intramuscularly with ASIS Device for 30 patients.
  Total cumulative Persistent % of Gadolinium intramuscularly on MRI at 6 hrs, 12 hrs, and 24 hrs.
  Other Names: Gadolinium Magnevist® (gadopentetate dimeglumine)
  Arms: Adductor pollicis; Biceps Brachii; Flexor Carpi Radialis; Flexor carpi ulnaris; Flexor digitorum profundus; Flexor digitorum sublimis; Flexor pollicis longus
Drug: Gadolinium — Gadolinium .1cc/ diluted with .9ccNS subdermally with ASIS Device for 30 patients.
  Total cumulative Persistent % of Gadolinium subdermally on MRI at 6 hrs, 12 hrs, and 24 hrs.
  Other Names: Gadolinium Magnevist® (gadopentetate dimeglumine)
  Arms: Adductor pollicis; Biceps Brachii; Flexor Carpi Radialis; Flexor carpi ulnaris; Flexor digitorum profundus; Flexor digitorum sublimis; Flexor pollicis longus
Drug: Gadolinium — Relative Prolongation Ability Score or total Persistent % of Gadolinium subdermally over total Persistent % of Gadolinium intramuscularly on MRI.
  Other Names: Gadolinium Magnevist® (gadopentetate dimeglumine)
  Arms: Adductor pollicis; Biceps Brachii; Flexor Carpi Radialis; Flexor carpi ulnaris; Flexor digitorum profundus; Flexor digitorum sublimis; Flexor pollicis longus
Drug: Efficacy of Botox intramuscularly at Week 6 — Efficacy of Botox intramuscularly at Week 6, in terms of Change from Baseline in PGAS, or improvement on the Physician Global Assessment Scale, and Change from Baseline in Elbow Ashworth, Change from Baseline in Wrist Ashworth, Change from Baseline in Finger Ashworth, and Change from Baseline in Thumb Ashworth.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change from Baseline in Elbow Ashworth; Change from Baseline in Finger Ashworth; Change from Baseline in PGAS; Change from Baseline in Thumb Ashworth; Change from Baseline in Wrist Ashworth
Drug: Efficacy of Botox intramuscularly at Week 12, — Efficacy of Botox intramuscularly at Week 12, in terms of Change from Baseline in PGAS, or improvement on the Physician Global Assessment Scale, and Change from Baseline in Elbow Ashworth, Change from Baseline in Wrist Ashworth, Change from Baseline in Finger Ashworth, and Change from Baseline in Thumb Ashworth.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change from Baseline in Elbow Ashworth; Change from Baseline in Finger Ashworth; Change from Baseline in PGAS; Change from Baseline in Thumb Ashworth; Change from Baseline in Wrist Ashworth
Drug: Efficacy of Botox intramuscularly at Week 18 — Efficacy of Botox intramuscularly at Week 18, in terms of Change from Baseline in PGAS, or improvement on the Physician Global Assessment Scale, and Change from Baseline in Elbow Ashworth, Change from Baseline in Wrist Ashworth, Change from Baseline in Finger Ashworth, and Change from Baseline in Thumb Ashworth.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change from Baseline in Elbow Ashworth; Change from Baseline in Finger Ashworth; Change from Baseline in PGAS; Change from Baseline in Thumb Ashworth; Change from Baseline in Wrist Ashworth
Drug: Efficacy of Botox intramuscularly at Week 24 — Efficacy of Botox intramuscularly at Week 24, in terms of Change from Baseline in PGAS, or improvement on the Physician Global Assessment Scale, and Change from Baseline in Elbow Ashworth, Change from Baseline in Wrist Ashworth, Change from Baseline in Finger Ashworth, and Change from Baseline in Thumb Ashworth.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change from Baseline in Elbow Ashworth; Change from Baseline in Finger Ashworth; Change from Baseline in PGAS; Change from Baseline in Thumb Ashworth; Change from Baseline in Wrist Ashworth
Drug: Efficacy of Botox intramuscularly at Week 30 — Efficacy of Botox intramuscularly at Week 30, in terms of Change from Baseline in PGAS, or improvement on the Physician Global Assessment Scale, and Change from Baseline in Elbow Ashworth, Change from Baseline in Wrist Ashworth, Change from Baseline in Finger Ashworth, and Change from Baseline in Thumb Ashworth.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change from Baseline in Elbow Ashworth; Change from Baseline in Finger Ashworth; Change from Baseline in PGAS; Change from Baseline in Thumb Ashworth; Change from Baseline in Wrist Ashworth
Drug: Efficacy of Botox subdermally at Week 6 — Efficacy of Botox subdermally at Week 6, in terms of Change from Baseline in PGAS, or improvement on the Physician Global Assessment Scale, and Change from Baseline in Elbow Ashworth, Change from Baseline in Wrist Ashworth, Change from Baseline in Finger Ashworth, and Change from Baseline in Thumb Ashworth.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change from Baseline in Elbow Ashworth; Change from Baseline in Finger Ashworth; Change from Baseline in PGAS; Change from Baseline in Thumb Ashworth; Change from Baseline in Wrist Ashworth
Drug: Efficacy of Botox subdermally at Week 12 — Efficacy of Botox subdermally at Week 12, in terms of Change from Baseline in PGAS, or improvement on the Physician Global Assessment Scale, and Change from Baseline in Elbow Ashworth, Change from Baseline in Wrist Ashworth, Change from Baseline in Finger Ashworth, and Change from Baseline in Thumb Ashworth.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change from Baseline in Elbow Ashworth; Change from Baseline in Finger Ashworth; Change from Baseline in PGAS; Change from Baseline in Thumb Ashworth; Change from Baseline in Wrist Ashworth
Drug: Efficacy of Botox subdermally at Week 18 — Efficacy of Botox subdermally at Week 18, in terms of Change from Baseline in PGAS, or improvement on the Physician Global Assessment Scale, and Change from Baseline in Elbow Ashworth, Change from Baseline in Wrist Ashworth, Change from Baseline in Finger Ashworth, and Change from Baseline in Thumb Ashworth.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change from Baseline in Elbow Ashworth; Change from Baseline in Finger Ashworth; Change from Baseline in PGAS; Change from Baseline in Thumb Ashworth; Change from Baseline in Wrist Ashworth
Drug: Efficacy of Botox subdermally at Week 24 — Efficacy of Botox subdermally at Week 24, in terms of Change from Baseline in PGAS, or improvement on the Physician Global Assessment Scale, and Change from Baseline in Elbow Ashworth, Change from Baseline in Wrist Ashworth, Change from Baseline in Finger Ashworth, and Change from Baseline in Thumb Ashworth.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change from Baseline in Elbow Ashworth; Change from Baseline in Finger Ashworth; Change from Baseline in PGAS; Change from Baseline in Thumb Ashworth; Change from Baseline in Wrist Ashworth
Drug: Efficacy of Botox subdermally at Week 30 — Efficacy of Botox subdermally at Week 30, in terms of Change from Baseline in PGAS, or improvement on the Physician Global Assessment Scale, and Change from Baseline in Elbow Ashworth, Change from Baseline in Wrist Ashworth, Change from Baseline in Finger Ashworth, and Change from Baseline in Thumb Ashworth.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change from Baseline in Elbow Ashworth; Change from Baseline in Finger Ashworth; Change from Baseline in PGAS; Change from Baseline in Thumb Ashworth; Change from Baseline in Wrist Ashworth
Drug: Adverse Reactions of Botox intramuscularly — Adverse Reactions of Botox (onabotulinumtoxinA) intramuscularly at Week 30, in number of Headache Migraine, Facial paresis, Eyelid ptosis, Bronchitis, Neck pain Musculoskeletal stiffness, Muscular weakness Myalgia, Musculoskeletal pain, Muscle spasms, Injection site pain, and Hypertension.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Adverse Reactions Injection site pain; Adverse Reactions with Bronchitis; Adverse Reactions with Eyelid ptosis; Adverse Reactions with Facial paresis; Adverse Reactions with Hypertension; Adverse Reactions with Muscle pain; Adverse Reactions with Muscle spasms; Adverse Reactions with Muscle stiffness; Adverse Reactions with Muscular weakness; Adverse Reactions with Myalgia; Adverse Reactions with Neck pain
Drug: Adverse Reactions of Botox subdermally — Adverse Reactions of Botox (onabotulinumtoxinA) subdermally at Week 30, in number of Headache Migraine, Facial paresis, Eyelid ptosis, Bronchitis, Neck pain Musculoskeletal stiffness, Muscular weakness Myalgia, Musculoskeletal pain, Muscle spasms, Injection site pain, and Hypertension.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Adverse Reactions Injection site pain; Adverse Reactions with Bronchitis; Adverse Reactions with Eyelid ptosis; Adverse Reactions with Facial paresis; Adverse Reactions with Hypertension; Adverse Reactions with Muscle pain; Adverse Reactions with Muscle spasms; Adverse Reactions with Muscle stiffness; Adverse Reactions with Muscular weakness; Adverse Reactions with Myalgia; Adverse Reactions with Neck pain

SUMMARY:
Botox act on nerve endings, yet there are no nerve endings inside the muscle, where they are typically injected. All nerves terminate on the fascia, where ASIS device can precisely deliver Botox by creating that subdermal bloodless space, between the skin and muscle. Thus enhancing and prolonging Botox's efficacy, at the same time prevent it's unnecessary adverse reactions and distant spread, especially since Botox has no reason to travel to the rest of the body any way.

DETAILED DESCRIPTION:
Aim 1 over 6 months will demonstrate ASIS device's consistent performance on 60 adult subjects with Upper limb Spasticity. Gadolinium will be injected with ASIS subdermally (30) or conventional intramuscularly (30) for these 7 muscle groups: Biceps Brachii, Flexor Carpi Radialis, Flexor Carpi Ulnaris, Flexor Digitorum Profundus, Flexor Digitorum Sublimis, Adductor Pollicis, and Flexor Pollicis Longus. An MRI will be taken promptly after Gadolinium injection, as starting reference, to which subsequent MRI taken at 6 hrs, 12 hrs, and 24 hrs later will be compared for Persistent %. Since there isn't a way to measure level of Gadolinium within it, or any other (e.g. Botox) for that matter, at least the Prolongation of Gadolinium may be approximated by the greater or longer Persistent % on MRI. However, this approximation can only work if the variables are minimized to the same population with Upper limb Spasticity, and these particular 7 muscle groups. Case in point, patients with Upper limb Spasticity presumably have hyperactivity in these 7 muscle groups, so expectantly will have shortened Gadolinium intramuscularly Persistent %, and somewhat reduced Gadolinium subdermally Persistent % as well due to agitation, thus these Persistent % values in Upper limb Spasticity patients will not be like those of normal patients, or even the same between these 7 different muscle groups. Therefore, the Relative Prolongation Ability Score or total Persistent % subdermally over total Persistent % intramuscularly, will be specific and valuable indicators to help us modify the Botox dosage and duration to inject into that "unknown" subdermal bloodless space for Aim 2.

Aim 2 over 12 months, using Botox, instead of Gadolinium, to demonstrate the advantages of ASIS device subdermally over intramuscularly, for the same 60 adult subjects with Upper limb Spasticity, on these particular 7 muscle groups: Biceps Brachii, Flexor Carpi Radialis, Flexor Carpi Ulnaris, Flexor Digitorum Profundus, Flexor Digitorum Sublimis, Adductor Pollicis, and Flexor Pollicis Longus. Hypothetically speaking, if that subdermal bloodless space in patients with e.g., Upper limb Spasticity somehow failed to show prolongation of half-life for Gadolinium in Aim 1, we can still proceed with primary interest being therapeutic comparison for Botox in Aim 2, in terms of improvement on the Physician Global Assessment Scale and Ashworth score (force required to move an extremity around a joint), at 6,12,18,24, and 30 weeks, and reduction in adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* Adults with history of stroke that resulted in a unilateral, upper-limb focal spasticity
* Wrist flexor tone of more than 2 and finger flexor tone of more than 2 as measured by the Ashworth Scale
* Ability to understand and follow verbal directions
* At least 1 functional disability item (hygiene, dressing, pain, or limb posture) with a rating of more than 2 on the Disability Assessment Scale (DAS)
* At least 1 functional task score at Day 0 that met the following criteria: nail filing less than 6, hand cleaning less than 6, holding a water bottle less than 4, brushing teeth less than 4, holding fruit (small, medium, or large equals no.

Exclusion Criteria:

* Stroke within 6 months of the study enrollment visit
* Females who are pregnant, nursing, or planning a pregnancy during the study period or who are not using a reliable means of contraception
* Previous or current Botox therapy of any type in the study limb
* Any medical condition that may put the patient at increased risk with Botox exposure or any other disorder that might have interfered with neuromuscular function
* Presence of fixed contracture of the study limb
* Limited use of the wrist and fingers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Relative Prolongation Ability Score for Gadolinium subdermally injected. | 6 months
  Gadolinium will be injected with ASIS subdermally (30) or intramuscularly (30) in Upper Limb Spasticity adult patients for these 7 muscle groups: Biceps Brachii, Flexor Carpi Radialis, Flexor Carpi Ulnaris, Flexor Digitorum Profundus, Flexor Digitorum Sublimis, Adductor Pollicis, and Flexor Pollicis Longus. MRI will be taken promptly after, as starting reference, to which subsequent MRI at 6 hrs, 12 hrs, and 24 hrs later will be compared for Persistent %. This approximation can only work if the variables are minimized to the same population with Upper Limb Spasticity, and these particular 7 muscle groups. The Relative Prolongation Ability Score or total Persistent % subdermally over total Persistent % intramuscularly, in Upper Limb Spasticity patients will not be same as normal patients, or even between these 7 different muscle groups, but valuable indicators to help us modify Botox dosage and duration to inject into "unknown" subdermal bloodless space for Aim 2.

SECONDARY OUTCOMES:
Efficacy of Botox intramuscularly vs. subdermally in Upper Limb Spasticity. | 12 months
  Efficacy of Botox intramuscularly vs. subdermally with ASIS Device at Week 6,12,18, 24, and 30; in terms of improvement on the Physician Global Assessment Scale (-4=very marked worsening to +4=very marked improvement). Also in terms of improvement, or Median Change from Baseline in Flexor Tone on Ashworth Scale, for Elbow, Wrist, Finger, and Thumb. Ashworth score (the force required to move an extremity around a joint):
  0 = No increase in muscle tone (none)
  1. = Slight increase in muscle tone, giving a 'catch' when the limb was flexed or extended (mild)
  2. = More marked increase in muscle tone but affected limb is easily flexed (moderate)
  3. = Considerable increase in muscle tone - passive movement difficult (severe)
  4. = Limb rigid in flexion or extension (very severe).

OTHER OUTCOMES:
Adverse Reactions of Botox intramuscularly vs. subdermally in Upper Limb Spasticity | 12 months
  Adverse Reactions of Botox intramuscularly vs. subdermally:
  Headache Migraine, Facial paresis, Eyelid ptosis, Bronchitis, Neck pain Musculoskeletal stiffness, Muscular weakness Myalgia, Musculoskeletal pain, Muscle spasms, Injection site pain, and Hypertension.

CONTACTS AND LOCATIONS:
Overall Officials: Li Nguyen, MD, Principal Investigator — AUTOMATIC SUBDERMAL INJECTOR SYSTEM INC; Thanh Phung,, MD, Principal Investigator — AUTOMATIC SUBDERMAL INJECTOR SYSTEM, INC
Locations (1):
- Automatic Subdermal Injector System, Inc, Westminster, California, United States

REFERENCES:
- [Background] Lorenc ZP, Kenkel JM, Fagien S, Hirmand H, Nestor MS, Sclafani AP, Sykes JM, Waldorf HA. A review of onabotulinumtoxinA (Botox). Aesthet Surg J. 2013 Mar;33(1 Suppl):9S-12S. doi: 10.1177/1090820X12474629. PMID 23515199
- [Background] Knopp MV, Balzer T, Esser M, Kashanian FK, Paul P, Niendorf HP. Assessment of utilization and pharmacovigilance based on spontaneous adverse event reporting of gadopentetate dimeglumine as a magnetic resonance contrast agent after 45 million administrations and 15 years of clinical use. Invest Radiol. 2006 Jun;41(6):491-9. doi: 10.1097/01.rli.0000209657.16115.42. PMID 16763467
- [Background] Turner-Stokes L, Ward A. Botulinum toxin in the management of spasticity in adults. Clin Med (Lond). 2002 Mar-Apr;2(2):128-30. doi: 10.7861/clinmedicine.2-2-128. PMID 11991094
- [Background] Patrick E, Ada L. The Tardieu Scale differentiates contracture from spasticity whereas the Ashworth Scale is confounded by it. Clin Rehabil. 2006 Feb;20(2):173-82. doi: 10.1191/0269215506cr922oa. PMID 16541938
- [Background] Jost WH, Hefter H, Reissig A, Kollewe K, Wissel J. Efficacy and safety of botulinum toxin type A (Dysport) for the treatment of post-stroke arm spasticity: results of the German-Austrian open-label post-marketing surveillance prospective study. J Neurol Sci. 2014 Feb 15;337(1-2):86-90. doi: 10.1016/j.jns.2013.11.022. Epub 2013 Nov 22. PMID 24361062
- [Background] Baker JA, Pereira G. The efficacy of Botulinum Toxin A for spasticity and pain in adults: a systematic review and meta-analysis using the Grades of Recommendation, Assessment, Development and Evaluation approach. Clin Rehabil. 2013 Dec;27(12):1084-96. doi: 10.1177/0269215513491274. Epub 2013 Jul 17. PMID 23864518
- [Background] Ghasemi M, Salari M, Khorvash F, Shaygannejad V. A literature review on the efficacy and safety of botulinum toxin: an injection in post-stroke spasticity. Int J Prev Med. 2013 May;4(Suppl 2):S147-58. PMID 23776717
- See also: Click here for more information about this study ASIS for Botox in Upper Limb Spasticity — http://www.asis-inc.com